CLINICAL TRIAL: NCT01828346
Title: A Phase 1b/2a, Open-label, Non-randomized Study of Birinapant in Combination With 5-azacitidine in Subjects With Myelodysplastic Syndrome Who Are Naïve, Refractory or Have Relapsed to 5-azacitidine Therapy
Brief Title: Birinapant With 5-azacitidine in MDS Subjects Who Are Naïve, Have Relapsed or Are Refractory to 5-azacitidine Therapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TetraLogic Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TL32711-0087
Record Dates: First submitted 2013-04-05; First posted 2013-04-10 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Myelodysplastic Syndrome
Keywords: TL32711; Birinapant; 5-Azacitidine; Myelodysplastic syndrome; MDS; Relapsed; Refractory; Failed; open-label; non-Randomized; dose-escalation; dose-expansion
MeSH Terms: conditions — Myelodysplastic Syndromes; Recurrence | interventions — birinapant; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): 5-Azacitidine plus birinapant
  Interventions: Drug: Birinapant; Drug: 5-Azacitidine

INTERVENTIONS:
Drug: Birinapant — Dose escalation part: (Drug escalation dose levels)
  * Dose Level (1) - 13mg/m2 (twice a week for 3 of 4 weeks)
  * Dose Level (-1) - 11 mg/m2 (twice a week for 3 of 4 weeks)
  * Dose Level (2) - 13mg/m2 (twice weekly x 4 weeks)
  * Dose Level (3a) - 17mg/m2 (twice weekly × 4 weeks)OR
  * Dose Level (3b) - 17mg/m2 (twice a week for 3 of 4 weeks)
  Other Names: TL32711
Drug: 5-Azacitidine — Dose Level (0) - 75mg/m2 daily
  Other Names: 5-AZA

SUMMARY:
This is a dose escalation followed by dose expansion study of TL32711 in combination with 5-Azacitidine in subjects with Myelodysplastic syndrome who are naïve, have relapsed or have failed prior 5-azacitidine therapy. Pre-clinical and mechanistic studies support that 5-Azacitidine may modulate pathways that enable birinapant-mediated anti-tumor activity.

DETAILED DESCRIPTION:
This is a Phase 1b/2a, open-label, non-randomized study in male and female subjects with MDS who are naïve, refractory or have relapsed to 5-Azacitidine therapy.

Primary Objective is to determine the maximum tolerated dose (MTD), recommended Phase 2 dose, and pharmacodynamics (PD) of birinapant (TL32711) when administered in combination with 5-azacitidine (5 AZA) in subjects with myelodysplastic syndrome (MDS) who are naïve, refractory or have relapsed to 5-AZA therapy.

Secondary Objectives are to determine the clinical activity using the International Working Group (IWG) (Cheson, 2006) Response Criteria for MDS during the Phase 1b dose escalation stage of the study and in the Phase 2a expansion cohort, to determine the pharmacokinetics (PK) of birinapant when administered with 5-AZA in plasma and to assess exploratory translational biomarkers of anti-tumor activity of birinapant in combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Men or women more than 18 years of age.
* Patients with high-risk Myelodysplastic Syndrome
* Performance status of greater or equal to 2 by the Eastern Cooperative Oncology Group (ECOG) scale.
* Subjects with high-risk MDS who are naïve to 5-Azacitidine or have previously received 5-AZA or decitabine as first-line cytotoxic therapy. Subjects with prior 5-Azacitidine therapy were evaluated to be either refractory or relapsed as determined by the Investigator, according to IWG response criteria.Subjects with relapsed or refractory disease may have only received prior 5-Azacitidine or decitabine.
* Hydroxyurea for patients with rapidly proliferative disease can be used up to 24 hours prior to therapy but not concomitantly with 5-Azacitidine.
* Adequate liver, pancreatic and renal function.
* Women of childbearing potential must have a negative serum pregnancy test at screening within 48 hours prior to the first dose
* Women of childbearing potential must agree to use 2 methods of adequate contraception

Exclusion Criteria:

* Subjects with life-threatening toxicity or non tolerability to prior 5-Azacitidine therapy.
* Subjects with hypoplastic Myelodysplastic syndrome.
* Subjects with >30% bone marrow blast cells.
* Subjects with malignant hepatic tumors or secondary malignancy within 2 years
* Known diagnosis of human immunodeficiency virus or chronic active Hepatitis B or C.
* Uncontrolled hypertension
* Impaired cardiac function, uncontrolled cardiac arrhythmias despite medications,
* QT interval corrected for heart rate (QTcB) more than 480 msec
* Lack of recovery of prior adverse events to Grade ≤1 severity (National Cancer Institute Common Terminology Criteria for Adverse Events version 4) (except alopecia) due to therapy administered prior to the initiation of study drug dosing.
* Nursing or pregnant women.
* Known allergy to any of the formulation components of birinapant.
* Known or suspected hypersensitivity to 5-Azacitidine or mannitol.
* Any concurrent disease and/or medical condition that, in the opinion of the Investigator, would prevent the subject's participation.
* History of Bell's Palsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-06; Primary Completion 2015-06 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gautam Borthakur, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (7):
- United States (7):
  - Palo Verde Hematology Oncology, Glendale, Arizona
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - California Cancer Associates for Research and Excellence, Fresno, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of Pennsylvania, Abramson Cancer Center, Philadelphia, Pennsylvania
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No